CLINICAL TRIAL: NCT02470780
Title: Treating Bacterial Overgrowth in Parkinson's Disease
Acronym: SIBO-PD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Alberto Espay, MD, MSc, Associate Professor of Neurology, University of Cincinnati
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-2175
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Parkinson's Disease; Small Intestinal Bacterial Overgrowth
MeSH Terms: conditions — Parkinson Disease | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Participants randomized to the drug ended their study participation at 3 months without switching over to a placebo. Those randomized to placebo were switched to the drug after 3 months and followed for another 3 months (6 months total).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Three-month follow-up (Experimental)
  Interventions: Drug: Rifaximin; Drug: Placebo
- Six-month follow-up (Experimental)
  Interventions: Drug: Rifaximin; Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin is an antibiotic used to treat SIBO. It is a 7-day course of treatment followed by three or six months of follow-up. This is a placebo-controlled study designed so that all participants will receive the active drug at least once during the study.
Drug: Placebo — Placebo matching Rifaximin treatment.

SUMMARY:
This study investigates the effect of treating Small Intestinal Bacterial Overgrowth (SIBO) in patients with Parkinson's Disease (PD). It will test the hypothesis that treating SIBO with the antibiotic rifaximin will improve motor complications in previously SIBO-positive PD patients.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) patients with motor fluctuations will be screened for the presence of Small Intestinal Bacterial Overgrowth (SIBO) using two hydrogen breath tests. SIBO-positive individuals will be eligible to enroll, and randomized to receive either rifaximin or placebo. This study includes two treatment regimens (including a placebo control), designed so that all patients will receive the active drug at some point during the trial. Motor outcomes will be followed for 3 or 6 months following enrollment, depending on the treatment arm to which the subject has been assigned. The primary endpoint is to assess the effect of rifaximin treatment to decrease "off" time in SIBO-positive PD patients.

This pilot study will support the design of a larger, randomized controlled trial investigating the effect of SIBO eradication on reducing motor complications in PD patients with motor fluctuations. The current proposal is designed to demonstrate our ability to detect and treat SIBO in PD patients with motor fluctuations, to inform selection of the best SIBO detection method, to determine the optimal timeline for assessing motor endpoints, and to estimate the duration of benefits after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* Daily "off" time ≥ 4 hours
* No changes in levodopa or any other dopaminergic medications expected during the course of the study
* Will be screened for cognitive ability (Montreal Cognitive Assessment score of ≥ 24) prior to enrollment
* Will be screened for presence of SIBO prior to enrollment

Exclusion Criteria:

* Any comorbid non-PD-associated gastrointestinal (e.g., achlorhydria) or systemic diseases that may alter absorption or confound the study results
* Exposure to proton pump inhibitors, immunosuppressive drugs, medications that affect GI motility (such as prokinetics, anticholinergics, and tricyclic antidepressants), antibiotics or any other drugs that affect the intestinal flora (such as laxatives) within a month prior to enrollment.
* Prior deep brain stimulation or ablative functional neurosurgery.
* Prior allergy to rifaximin
* Women who are pregnant, lactating, or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rifaximin (3-month Follow-up): Participants in this group received a 7-day treatment with Rifaximin and were followed for three months. Participants were blinded to their treatment assignment until the conclusions of the 3-month visit.
- Placebo Then Rifaximin (6-month Follow-up): Participants in this group received a 7-day treatment with placebo and were followed for three months. Participants were blinded to their treatment assignment until the conclusions of the 3-month visit. At the end of the 3-month visit, they were given a 7-day course of Rifaximin and followed for an additional 3 months.
Period: Phase 1
Arm/Group | Rifaximin (3-month Follow-up) | Placebo Then Rifaximin (6-month Follow-up)
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | Rifaximin (3-month Follow-up) | Placebo Then Rifaximin (6-month Follow-up)
Started | 0 (Participants in this arm completed the study in 3 months after the first phase.) | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin (3-month Follow-up) | Placebo Then Rifaximin (6-month Follow-up) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (5.3) | 61.2 (5.8) | 66.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
OFF time [Mean (Standard Deviation); unit: hours] — OFF time is the time levodopa isn't effective and symptoms of Parkinson's disease reemerge.
  hours | 1.4 (2.0) | 5.2 (0.7) | 3.3 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in "Off" Time as Measured by Patient Diary
Description: OFF time is the time in which levodopa has ceased to be effective and Parkinsonian symptoms reemerge.
Time Frame: baseline to 1 month and 3 months; new baseline at 3 months to 4 months and 6 months
Population: Participants in this group completed the study at 3 months after treatment with rifaximin. They were not assessed at 4 and 6 months.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Placebo Then Rifaximin: Participants in this group received a 7-day treatment with placebo and then received rifaximin.
Arm/Group | Rifaximin (3-month Follow-up) | Placebo Then Rifaximin
Number analyzed (Participants) | 2 | 2
hours
  1 month change from baseline | -1.4 (2.0) | -2.8 (0.7)
  3 month change from baseline | -0.9 (1.3) | -2.0 (2.8)
  4 month change from new baseline (P to R group only): number analyzed (Participants) | 0 | 2
  4 month change from new baseline (P to R group only) |  | -1.4 (2.5)
  6 month change from new baseline (P to R group only): number analyzed (Participants) | 0 | 2
  6 month change from new baseline (P to R group only) |  | -2.2 (3.5)

2. Primary Outcome: Change in "Off" Time as Measured by Wireless Computer Monitoring System
Description: This outcome measure was not analyzed due to low subject enrollment as well as poor subject compliance or data quality in some cases.
Time Frame: 1, 3, and 6 months
Population: This outcome measure was not analyzed due to low subject enrollment as well as poor subject compliance or data quality in some cases. No data were collected for this outcome measure.
Groups:
- Placebo Then Rifaximin (6-month Follow-up: Participants in this group received a 7-day treatment with placebo and were followed for three months. Participants were blinded to their treatment assignment until the conclusions of the 3-month visit. At the end of the 3-month visit, they were given a 7-day course of Rifaximin and followed for an additional 3 months.
Arm/Group | Rifaximin (3-month Follow-up) | Placebo Then Rifaximin (6-month Follow-up
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During enrollment period (3 months or 6 months, depending on group assignment)
Description: Adverse events related to disease state or disease progression were not collected. Only adverse events related to study interventions were collected.
Groups:
- Rifaximin: Participants in this group received a 7-day treatment with Rifaximin and were followed for three months. Participants were blinded to their treatment assignment until the conclusions of the 3-month visit.
- Placebo: Participants in this group received a 7-day treatment with placebo and were followed for three months.
Arm/Group | Rifaximin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02470780/Prot_SAP_000.pdf